CLINICAL TRIAL: NCT00185692
Title: Allogeneic Hematopoietic Cell Transplantation of Positively Selected CD34+ Cells and Defined Inoculum of T Cells From Related Haploidentical Donors for Older Patients With Indolent Hematologic Malignancies
Brief Title: Allogeneic Transplantation From Related Haploidentical Donors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robert Lowsky, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13371; 75117 (Other: Stanford University Alternate IRB Approval Number); BMT124 (Other: OnCore)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2017-01-26 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2015-01

CONDITIONS: Blood Cancer; Leukemia; Graft Versus Host Disease; Malignancy; CLL; NHL; Hodgkin's Disease; MDS
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Graft vs Host Disease; Neoplasms; Hodgkin Disease | interventions — Peripheral Blood Stem Cell Transplantation; Antilymphocyte Serum; Cyclosporine; Mycophenolic Acid; Granulocyte Colony-Stimulating Factor; Methylprednisolone Hemisuccinate; Methylprednisolone; Methylprednisolone Acetate; Acetaminophen; aminophylline, cycloclenbutrerol, diphenydramine, phenobarbital drug combination; Diphenhydramine; Hydrocortisone; hydrocortisone sodium phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplantation of CD34+ cells (Experimental): Week #1: Total Lymphoid Inrradiation (TLI) 120 cGy + Anti-thymocyte Globulin (ATG) 1.5 mg/kg + Solumedrol 1.0 mg/kg Daily for 5 days.
  Week #2: TLI 120 cGy (3 days a week, double on the 4th day) 5 days of CSP (oraly) one day after TLI was started. 3 days of MMF 4 days after TLI was started.
  Interventions: Procedure: non-myeloablative hematopoietic cell transplantation; Drug: Anti-Thymocyte Globulin; Drug: Cyclosporine; Drug: Mycophenolate Mofetil; Drug: G-CSF; Drug: Solumedrol; Drug: Acetaminophen; Drug: Diphenydramine; Drug: Hydrocortisone

INTERVENTIONS:
Procedure: non-myeloablative hematopoietic cell transplantation — TLI and ATG infusion of the donor graft Post-transplant immunosuppression with cyclosporine and mycophenolate mofetil.
  Other Names: Peripheral-blood stem-cell transplantation
Drug: Anti-Thymocyte Globulin — 1.5 mg/kg QD x 5, IV. Dosage will be based on body weight. Purified, sterile IgG fraction of immune serum of rabbits immumixied with human thymus lymphocyte. This drug acts to modify the number and function of lymphocytes.
  Other Names: ATG
Drug: Cyclosporine — 6.25 mg/kg BID, PO.Mechanism of action is inhibition of T-cell activation by binding to a cytoplasmic protein (cyclophillin).
  Other Names: INN/BAN; USAN; CSA
Drug: Mycophenolate Mofetil — 15 mg/kg Q 8 hours, PO. Inhibtis the enzme inosine monophsophate dehydrogenase (MPDII) noncompetitively which blocks the de nobo synthesis of guanosine required for DNA synthesis and has an effect on T and B cells.
  Other Names: MMF; CellCept
Drug: G-CSF — 16 mg/kg, SQ Growth factor used to make bone marrow produce more blood cells
  Other Names: Granulocyte colony-stimulating factor; CSF 3
Drug: Solumedrol — 1.0 mg/kg IV 2 hours prior to ATG Used to treat severe inflamation
  Other Names: 6-Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Sodium Succinate
Drug: Acetaminophen — 650 mg PO, 30 minutes prior to infusion Pain reliever
  Other Names: Tylenol
Drug: Diphenydramine — 50 mg IV, 30 minutes prior to infusion Used to relieve allergy symptoms
  Other Names: Benadryl; Allermax; Q-Dryl; Diphen Cough
Drug: Hydrocortisone — 100 mg IV, 1 hour prior to infusion Used to relieve itching, redness and swelling of the skin
  Other Names: Hydrocortisone Sodium Phosphate

SUMMARY:
The purpose of the study is to evaluate the feasibility and safety of transplanting CD34+ selected hematopoietic cells from a haploidentical related donor following a nonmyeloablative regimen of total lymphoid irradiation (TLI) and antithymocyte globulin (ATG).

DETAILED DESCRIPTION:
An alternative to conventional allogeneic bone marrow transplantation is by using a non-myeloablative conditioning regimen. This regime would consist of both; total lymphoid irradiation (TLI) and anti-thymocyte globulin (ATG). Used in combination to achieve engraftment of haploidentical CD34+ selected peripheral blood stem cells in older patients or patients with underlying medical conditions that preclude standard allogeneic treatment. The expected results of this transplant regime will be expected to result in hematopoietic and immunologic reconstitution, decreased deaths related to the treatment regimen and decreased gravft-vs-host disease (GVHD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years with hematologic malignancies treatable by a mixed chimera allogeneic HCT.
* For patients ≤ 50 years of age with hematologic malignacies treatable with mixed chimera HCT who because of pre-exisiting medical conditions or prior therapy are considered to be at high risk for regimen-related toxicity associated with conventional transplants.
* Indolent advanced stage NHL, CLL, HD - Must have received and failed front-line therapy.
* Multiple myeloma (Stage II or III) - Must have received prior chemotherapy. Consolidation after prior autografting is permitted.
* AML/ALL - Must be in complete hematologic remission and have received cytotoxic chemotherapy at some stage before transplant. Patients with molecular or cytogenetic relapse will be accepted providing a donor is available. Patients with persistent or refractory disease will be considered on a case by case basis and transplants must be approved by the principal investigator.
* CML - Patients will be accepted in chronic or accelerated phase. Patients who have received prior autografts after high dose therapy or have undergone intensive chemotherapy for either peripheral blood stem cell mobilization or treatment of advanced CML may be enrolled provided they are in CR, chronic phase or accelerated phase.
* MDS - All patients with MDS will be eligible for this protocol, however, those patients with >10% blasts will require chemotherapy to reduce the blast % to < 10%.
* SAA - Patients with severe aplastic anemia who have failed front line therapy.
* A fully HLA-identical sibling donor is not available.
* A matched unrelated donor has not been identified.
* A haploidentical related donor is available who is in good health and does not have contraindications to donation.

Exclusion Criteria:

* Patients with rapidly progressive intermediate or high grade NHL
* Uncontrolled CNS involvement with disease
* Fertile men
* Women unwilling to use contraceptive techniques during and for 12 months following treatment
* Females who are pregnant
* Cardiac function: ejection fraction < 30% or cardiac failure requiring therapy
* Pulmonary: DLCO < 40% predicted and/or receiving supplementary continuous oxygen
* Liver function abnormalities: elevation of bilirubin to > 4 mg/dl and/or transaminases > 3x the upper limit of normal. If hyperbilirubinemai is due to a known cause that will not increase the risks of transplant, than this upper limit may be exceeded.
* Renal: creatinine clearance < 50 cc/min (24 hour urine collection)
* Karnofsky performance score < 60%
* Patients with poorly controlled hypertension.
* Documented fungal disease that persists despite treatment
* HIV positive patients.
* Hepatitis B and C positive patients will be evaluated on a case by case basis
* Psychiatric disorders or psychosocial problems which in the opinion of the primary physician or principal investigator would place the patient at unacceptable risk from this regimen.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2000-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lowsky, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transplating of CD34+ Selected Hematopietic Cells
Started | 16
Completed | 0
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Transplating of CD34+ Selected Hematopietic Cells
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 52 [14 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Engraftment of Haploidentical CD34+ Selected Blood Stem Cells in Older Patients or Those With Medical Co-morbidities Following Total Lymphoid Irradiation and Antithymocyte Globulin Transplant Conditioning
Description: number achieving donor cell engraftment (>95%) by day 90 after transplant.
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Groups:
- Transplantation of CD34+ Cells: Week #1: Total Lymphoid Inrradiation (TLI) 120 cGy + Anti-thymocyte Globulin (ATG) 1.5 mg/kg + Solumedrol 1.0 mg/kg Daily for 5 days.
  Week #2: TLI 120 cGy (3 days a week, double on the 4th day) 5 days of CSP (oraly) one day after TLI was started. 3 days of MMF 4 days after TLI was started.
  non-myeloablative hematopoietic cell transplantation: TLI and ATG infusion of the donor graft Post-transplant immunosuppression with cyclosporine and mycophenolate mofetil.
  Anti-Thymocyte Globulin: 1.5 mg/kg QD x 5, IV. Dosage will be based on body weight.
  Purified, sterile IgG fraction of immune serum of rabbits immumixied with human thymus lymphocyte. This drug acts to modify the number and function of lymphocytes.
  Cyclosporine: 6.25 mg/kg BID, PO.Mechanism of action is inhibition of T-cell activation by binding to a cytoplasmic protein (cyclophillin).
  Mycophenolate Mofetil: 15 mg/kg Q 8 hours, PO. Inhibtis the enzme inosine monophsophate dehydrogenase (MPDII) noncompetitively
Arm/Group | Transplantation of CD34+ Cells
Number analyzed (Participants) | 16
Participants | 4

2. Secondary Outcome: Acute Graft-versus-Host Disease (GVHD) Grade 2-4 Risk From Time of Transplant Until Day 90 Post-transplant
Description: GVHD grading system goes from 0-4 where grade 4 is the most severe. Grade 0 and 1 do not require systemic treatment, Grade 2-4 require treatment. This trial evaluated the risk of developing acute GVHD grades 2-4 within 90 days of transplant.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Transplantation of CD34+ Cells
Number analyzed (Participants) | 16
Participants | 1

ADVERSE EVENTS:
Time Frame: 120 days
Description: Non-serious adverse events were not collected.
Arm/Group | CD34+ Selected Hematopietic Cells
Serious Adverse Events (participants affected / at risk) | 14/16
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD34+ Selected Hematopietic Cells (N=16)
Death (General disorders) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes